CLINICAL TRIAL: NCT03557853
Title: A Prospective Observational Study to Evaluate Clinical and Radiological Manifestations of Coxitis in Patients With Ankylosing Spondylitis Treated With Simponi® (Golimumab)
Brief Title: Clinical and Radiological Manifestations of Coxitis in Patients With Ankylosing Spondylitis Treated With Golimumab
Acronym: GO-COX
Status: Completed | Type: Observational
Sponsor: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MK-8259-021
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-03

CONDITIONS: Ankylosing Spondylitis; Coxitis
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — golimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Golimumab injection: Patients with ankylosing spondylitis and coxitis being treated with Simponi (golimumab) according to local clinical practice and label.
  Interventions: Drug: Golimumab Injection

INTERVENTIONS:
Drug: Golimumab Injection — Simponi (golimumab) in fixed dose of 50 mg sc per month according to local label and local clinical practice.
  Other Names: Based on decision of investigators.

SUMMARY:
Rationale. Coxitis in AS is inflammation of hip(s) affecting significant number of patients. It is associated with worse function and more expressed axial disease requiring hip replacement at end-stage. Number of studies dedicated to coxitis treated with TNF alpha inhibitors is very limited.

Primary objective. To evaluate change of functional impairment in AS patients with coxitis from baseline to 12 months of therapy with golimumab by BASFI in daily clinical practice

Study design. This study is a non-interventional prospective observational cohort study conducted in multiple centers across Russia.

Study population. Patients with ankylosing spondylitis (according to the modified New York criteria) with coxitis newly prescribed golimumab during the course of usual clinical care will be enrolled and followed prospectively for 24 months with data collection at the approximate time points: baseline (pre-treatment) and consequent every 6 months. Patients will receive golimumab as prescribed in regular clinical practice.

Statistical Methods. Quantitative variables will be tested for normal distribution using the Shapiro-Wilk test. The hypothesis of equality of variances will be tested using Levene's test. Quantitative variables matching a normal distribution will be described in terms of the mean ± standard deviation, and values outside of the normal distribution as medians, 25% and 75% quartiles. Qualitative variables will be presented in the form of percentages of the absolute value N.

Sample Size and Power Calculations. Sample size calculation is based on data from GO-RAISE registration study in which golimumab was evaluated in patients with AS. The baseline BASFI was 5.0 which changed by mean (± SD, standard deviation) -2.5 (± 2.12) at week 52 (approximately 12 months). The analysis of the data shows that the minimum necessary sample size should be 18 patients to show a statistically significant change of BASFI from baseline to 12 months. On this basis and considering that the dropout rate over the two years is expected to be 30%, we decided that the necessary number of patients to be included into protocol should be 39 individuals. It is expected that around 27 patients will be included in the patient set completing the study. Power of the study is 90% with formula evaluation P = 1-β where P is power and β is type 2 error = 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years of age) with definite AS (as per modified New York criteria)
2. Coxitis with BASRI-hip score 0-2
3. Newly prescribed golimumab according to usual clinical practice
4. Naïve to anti-TNFs or other biologic agents prior to initiation of golimumab as indicated by the patient's medical records
5. Patient is enrolled after the investigator's decision to treat with golimumab, but before initiation of treatment with golimumab
6. Patient was informed of the benefits and risks of golimumab as per normal practice using the product leaflet
7. Signed informed consent form

Exclusion Criteria:

1. Any contraindication to golimumab in accordance to the label of Simponi®
2. BASRI-hip score 3-4
3. Any contraindication to MRI, e.g. previous hip joint replacement, heart pace maker.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ankylosing spondylitis and coxitis followed in normal practice, in whom golimumab has been newly prescribed.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Lukyanova, MD, Study Director — MSD Pharmaceuticals LLC
Locations (6):
- Russia (6):
  - KhMAO Regional Clinical Hospital, Khanty-Mansiysk
  - Moscow Clinical Scientific Center, Moscow
  - Pirogov National Medical Surgical Center, Moscow
  - Rheumatology Research Institute, Moscow
  - Regional Clinical Hospital #2, Rostov-on-Don
  - City Clinical Hospital, Yakutsk

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At least 18 patients to be recruited and followed-up for 12 months for preliminary statistical analysis based on the primary end-point (change of BASFI in 12 months after baseline).
Period: 12 Months of Follow-up: Interim Analysis
Arm/Group | Golimumab Injection
Started | 39
Completed (22 patients completed 12 months of follow-up and entered into the preliminary statistical analysis.) | 22
Not Completed | 17
Period: 24 Weeks of Follow-up: Final Analysis
Arm/Group | Golimumab Injection
Started | 39
Completed | 30
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.21 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 39
Coxitis symptoms duration [Median (Full Range); unit: months] | 24 [1 to 170]
Bath Ankylosing Spondylitis Functionality Index (BASFI) [Median (Inter-Quartile Range); unit: units on a scale] — The BASFI is a self-assessment instrument for defining functional ability in patients with AS. Contains 10 items: 8 items concerning activities referring to the functional anatomy of the patients (bending, reaching, changing position, standing, turning, and climbing steps) and 2 items assessing the patients' ability to cope with everyday life. Consists of Numeric response scale (0-10) from "easy" to "impossible." The mean of the 10 individual scales (scores) gives the BASFI score - a value between 0 and 10 with 0 reflecting no functional impairments and 10 reflecting maximal impairment. Population: Results of clinical effect assessment population are presented (n=30)
  units on a scale
    number analyzed (Participants) | 30
    (all) | 3.9 [1.7 to 5.6]
Bath Ankylosing Spondylitis Metrological Index (BASMI) [Median (Inter-Quartile Range); unit: units on a scale] — The Bath Ankylosing Spondylitis Metrology Index (BASMI) is used to assess mobility of spine and hip joints. The BASMI score is a sum of the 5 measures: cervical rotation (>85.0° to ≤8.5°), tragus to wall distance (<10 cm to ≥38 cm), lumbar flexion (>7.0 cm to ≤0.7 cm), lumbar side flexion (>20.0 cm to <1.2 cm), and intermalleolar distance (≥120 cm to <30 cm). Each item is scored from 0 to 10 based on deﬁned cut points. The scale of the BASMI ranges from 0 to 10, where 0 is no mobility limitation and 10 is a very severe limitation. Population: Results of clinical effect assessment population are presented (n=30)
  units on a scale
    number analyzed (Participants) | 30
    (all) | 3.0 [1.0 to 4.0]
Ankylosing Spondylitis Disease Activity Score (ASDAS-CRP) [Median (Inter-Quartile Range); unit: units on a scale] — The ASDAS-CRP is to measure disease activity based on a composite score. The score includes patient-reported assessments of back pain, duration of morning stiffness, peripheral joint pain and/or swelling, general well-being, and a serologic marker of inflammation C-reactive protein (CRP). Patient response items and a serologic measure of inflammation are mathematically combined to give the ASDAS-CRP. Score ranges from zero (reflecting no disease activity) with the upper end of the scale being determined by the level of the CRP. Population: Results of clinical effect assessment population are presented (n=30)
  units on a scale
    number analyzed (Participants) | 30
    (all) | 3.5 [2.7 to 4.3]
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) [Median (Inter-Quartile Range); unit: units on a scale] — The BASDAI is an instrument to measure disease activity in AS based on a composite score.The index includes patient-reported levels of back pain, fatigue, peripheral joint pain and swelling, localized tenderness, and the duration and severity of morning stiffness. It contains 6 items with numeric response scales (0-10) or visual analog scales (VAS, 0-10 cm) anchored by adjectival descriptors "none" and "very severe." Duration of morning stiffness is anchored by a time scale (0-2 or more hours). Population: Results of clinical effect assessment population are presented (n=30)
  units on a scale
    number analyzed (Participants) | 30
    (all) | 4.6 [3.4 to 6.1]
Bath Ankylosing Spondylitis Radiographic Score (BASRI) Right Hip [Median (Inter-Quartile Range); unit: units on a scale] — The BASRI-hip is a score of structural impairment of hip on X-ray images:
  0 - no change; 1 - suspicious: focal joint space narrowing; 2 - mild: circumferential joint space narrowing >2mm; 3 - moderate: circumferential joint space narrowing ≤ 2mm or bone-on-bone apposition of <2 cm; 4 - severe: bone deformity or bone-on-bone apposition of ≥2 cm. Population: Results of clinical effect assessment population are presented (n=30)
  units on a scale
    number analyzed (Participants) | 30
    (all) | 1.0 [1.0 to 2.0]
Bath Ankylosing Spondylitis Radiographic Score (BASRI) Left Hip [Median (Inter-Quartile Range); unit: units on a scale] — The BASRI-hip is a score of structural impairment of hip on X-ray images:
  0 - no change; 1 - suspicious: focal joint space narrowing; 2 - mild: circumferential joint space narrowing >2mm; 3 - moderate: circumferential joint space narrowing ≤ 2mm or bone-on-bone apposition of <2 cm; 4 - severe: bone deformity or bone-on-bone apposition of ≥2 cm. Population: Results of clinical effect assessment population are presented (n=30)
  units on a scale
    number analyzed (Participants) | 30
    (all) | 1.0 [1.0 to 2.0]
Percentage of participants without MRI Inflammatory Lesions [Count of Participants; unit: Participants] — There were no formal scores for MRI of hips at time of study initiation. Information on hips MRI (STIR (short tau inversion recovery) sequence and fat-saturated contrast-enhanced T1-weighted sequence) were collected based on availability: No lesions suggesting inflammation; Subchondral bone marrow edema (expressed as Yes or No); Joint effusion (expressed as Yes or No); Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No); Fatty degeneration (expressed as Yes or No). Population: Data are based on available MRI results suitable for paired analysis.
  Participants
    Right Hip: number analyzed (Participants) | 19
    Right Hip | 4
    Left Hip: number analyzed (Participants) | 19
    Left Hip | 3
Percentage of patients without Hips US Inflammatory Lesions [Count of Participants; unit: Participants] — There were no standardized US scores available for hips at the time of study initiation. Information on hip(s) US was collected for patients based on availability in the patient charts: Joint effusion (expressed as Yes or No); Distance between lower margin of femoral neck and lower part of joint capsule expressed in millimeters; Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No). Population: Data are based on available US results suitable for paired analysis.
  Participants
    Right Hip: number analyzed (Participants) | 21
    Right Hip | 3
    Left Hip: number analyzed (Participants) | 21
    Left Hip | 3

OUTCOME MEASURES:

1. Primary Outcome: BASFI (Bath Ankylosing Spodylitis Functionality Index) at 12 Months of Follow-up
Description: The BASFI is a self-assessment instrument for defining functional ability in patients with AS. Contains 10 items: 8 items concerning activities referring to the functional anatomy of the patients (bending, reaching, changing position, standing, turning, and climbing steps) and 2 items assessing the patients' ability to cope with everyday life. Consists of Numeric response scale (0-10) from "easy" to "impossible." The mean of the 10 individual scales (scores) gives the BASFI score - a value between 0 and 10 with 0 reflecting no functional impairments and 10 reflecting maximal impairment.
Time Frame: From baseline to 12 months
Population: Patients completed 12 months follow-up from the baseline. Results of clinical effect assessment population are presented (n=30)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.0 [0.0 to 2.7]

2. Secondary Outcome: BASFI (Bath Ankylosing Spodylitis Functionality Index) at 24 Months of Follow-up
Description: as for outcome 1
Time Frame: From baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.1 [0.0 to 2.7]

3. Secondary Outcome: BASMI (Bath Ankylosing Spodylitis Mobility Index) at 12 Months of Follow-up
Description: The Bath Ankylosing Spondylitis Metrology Index (BASMI) is used to assess mobility of spine and hip joints. The BASMI score is a sum of the 5 measures: cervical rotation (>85.0° to ≤8.5°), tragus to wall distance (<10 cm to ≥38 cm), lumbar flexion (>7.0 cm to ≤0.7 cm), lumbar side flexion (>20.0 cm to <1.2 cm), and intermalleolar distance (≥120 cm to <30 cm). Each item is scored from 0 to 10 based on deﬁned cut points. The scale of the BASMI ranges from 0 to 10, where 0 is no mobility limitation and 10 is a very severe limitation.
Time Frame: From baseline to 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.0 [0.0 to 2.0]

4. Secondary Outcome: BASMI (Bath Ankylosing Spodylitis Mobility Index) at 24 Months of Follow-up
Description: as for outcome 3
Time Frame: From baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 0.5 [0.0 to 2.0]

5. Secondary Outcome: ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score) at 12 Months of Follow-up
Description: The ASDAS-CRP is to measure disease activity based on a composite score. The score includes patient-reported assessments of back pain, duration of morning stiffness, peripheral joint pain and/or swelling, general well-being, and a serologic marker of inflammation C-reactive protein (CRP). Patient response items and a serologic measure of inflammation are mathematically combined to give the ASDAS-CRP. Score ranges from zero (reflecting no disease activity) with the upper end of the scale being determined by the level of the CRP.
Time Frame: From baseline to 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.3 [1.0 to 1.9]

6. Secondary Outcome: ASDAS-CRP (Ankylosing Spondylitis Disease Activity Score) at 24 Months of Follow-up
Description: as for outcome 5
Time Frame: From baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.1 [0.9 to 1.7]

7. Secondary Outcome: BASDAI (Bath AS Disease Activity Index) at 12 Months of Follow-up
Description: The BASDAI is an instrument to measure disease activity in AS based on a composite score.The index includes patient-reported levels of back pain, fatigue, peripheral joint pain and swelling, localized tenderness, and the duration and severity of morning stiffness. It contains 6 items with numeric response scales (0-10) or visual analog scales (VAS, 0-10 cm) anchored by adjectival descriptors "none" and "very severe." Duration of morning stiffness is anchored by a time scale (0-2 or more hours).
Time Frame: From baseline to 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.0 [0.6 to 2.9]

8. Secondary Outcome: BASDAI (Bath AS Disease Activity Index) at 24 Months of Follow-up
Description: as for outcome 7
Time Frame: From baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale | 1.1 [0.2 to 3.0]

9. Secondary Outcome: BASRI-hip (Bath Ankylosing Spondylitis Radiology Index) at 12 Months of Follow-up
Description: The BASRI-hip is a score of structural impairment of hip on X-ray images:
  0 - no change; 1 - suspicious: focal joint space narrowing; 2 - mild: circumferential joint space narrowing >2mm; 3 - moderate: circumferential joint space narrowing ≤ 2mm or bone-on-bone apposition of <2 cm; 4 - severe: bone deformity or bone-on-bone apposition of ≥2 cm.
Time Frame: From baseline to 12 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale
  Right Hip | 1.0 [1.0 to 2.0]
  Left Hip | 1.0 [1.0 to 2.0]

10. Secondary Outcome: BASRI-hip (Bath Ankylosing Spondylitis Radiology Index) at 24 Months of Follow-up
Description: as for outcome 9
Time Frame: From baseline to 24 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 30
units on a scale
  Right Hip | 1.0 [1.0 to 2.0]
  Left Hip | 2.0 [1.0 to 2.0]

11. Other Pre Specified Outcome: Percentage of Participants Without MRI Inflammatory Lesions in the Right Hip at 6 Months of Follow-up
Description: Percentage of participants without MRI Inflammatory Lesions in the Right Hip at 6 months of follow-up based on result available and suitable for paired analysis.
  There were no formal scores for MRI of hips at time of study initiation. Information on hips MRI (STIR (short tau inversion recovery) sequence and fat-saturated contrast-enhanced T1-weighted sequence) were collected based on availability: No lesions suggesting inflammation; Subchondral bone marrow edema (expressed as Yes or No); Joint effusion (expressed as Yes or No); Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No); Fatty degeneration (expressed as Yes or No).
Time Frame: 6 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 19
Participants | 7

12. Other Pre Specified Outcome: Percentage of Participants Without MRI Inflammatory Lesions in the Left Hip at 6 Months of Follow-up
Description: Percentage of participants without MRI Inflammatory Lesions in the Left Hip at 6 months of follow-up based on result available and suitable for paired analysis.
  There were no formal scores for MRI of hips at time of study initiation. Information on hips MRI (STIR (short tau inversion recovery) sequence and fat-saturated contrast-enhanced T1-weighted sequence) were collected based on availability: No lesions suggesting inflammation; Subchondral bone marrow edema (expressed as Yes or No); Joint effusion (expressed as Yes or No); Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No); Fatty degeneration (expressed as Yes or No).
Time Frame: 6 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 19
Participants | 6

13. Other Pre Specified Outcome: Percentage of Participants Without MRI Inflammatory Lesions in the Right Hip at 12 Months of Follow-up
Description: Percentage of participants without MRI Inflammatory Lesions in the Right Hip at 12 months of follow-up based on result available and suitable for paired analysis.
  There were no formal scores for MRI of hips at time of study initiation. Information on hips MRI (STIR (short tau inversion recovery) sequence and fat-saturated contrast-enhanced T1-weighted sequence) were collected based on availability: No lesions suggesting inflammation; Subchondral bone marrow edema (expressed as Yes or No); Joint effusion (expressed as Yes or No); Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No); Fatty degeneration (expressed as Yes or No).
Time Frame: 12 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 13
Participants | 8

14. Other Pre Specified Outcome: Percentage of Participants Without MRI Inflammatory Lesions in the Left Hip at 12 Months of Follow-up
Description: Percentage of participants without MRI Inflammatory Lesions in the Left Hip at 12 months of follow-up based on result available and suitable for paired analysis.
  There were no formal scores for MRI of hips at time of study initiation. Information on hips MRI (STIR (short tau inversion recovery) sequence and fat-saturated contrast-enhanced T1-weighted sequence) were collected based on availability: No lesions suggesting inflammation; Subchondral bone marrow edema (expressed as Yes or No); Joint effusion (expressed as Yes or No); Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No); Fatty degeneration (expressed as Yes or No).
Time Frame: 12 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 13
Participants | 5

15. Other Pre Specified Outcome: Percentage of Participants Without US Inflammatory Lesions in the Right Hip at 6 Months of Follow-up
Description: Percentage of participants without US Inflammatory Lesions in the Right Hip at 6 months of follow-up based on result available and suitable for paired analysis.
  There were no standardized US scores available for hips at the time of study initiation. Information on hip(s) US was collected for patients based on availability in the patient charts: Joint effusion (expressed as Yes or No); Distance between lower margin of femoral neck and lower part of joint capsule expressed in millimeters; Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No).
Time Frame: 6 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 21
Participants | 11

16. Other Pre Specified Outcome: Percentage of Participants Without US Inflammatory Lesions in the Left Hip at 6 Months of Follow-up
Description: Percentage of participants without US Inflammatory Lesions in the Left Hip at 6 months of follow-up based on result available and suitable for paired analysis.
  There were no standardized US scores available for hips at the time of study initiation. Information on hip(s) US was collected for patients based on availability in the patient charts: Joint effusion (expressed as Yes or No); Distance between lower margin of femoral neck and lower part of joint capsule expressed in millimeters; Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No).
Time Frame: 6 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 21
Participants | 9

17. Other Pre Specified Outcome: Percentage of Participants Without US Inflammatory Lesions in the Right Hip at 12 Months of Follow-up
Description: Percentage of participants without US Inflammatory Lesions in the Right Hip at 12 months of follow-up based on result available and suitable for paired analysis.
  There were no standardized US scores available for hips at the time of study initiation. Information on hip(s) US was collected for patients based on availability in the patient charts: Joint effusion (expressed as Yes or No); Distance between lower margin of femoral neck and lower part of joint capsule expressed in millimeters; Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No).
Time Frame: 12 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 18
Participants | 8

18. Other Pre Specified Outcome: Percentage of Participants Without US Inflammatory Lesions in the Left Hip at 12 Months of Follow-up
Description: Percentage of participants without US Inflammatory Lesions in the Left Hip at 12 months of follow-up based on result available and suitable for paired analysis.
  There were no standardized US scores available for hips at the time of study initiation. Information on hip(s) US was collected for patients based on availability in the patient charts: Joint effusion (expressed as Yes or No); Distance between lower margin of femoral neck and lower part of joint capsule expressed in millimeters; Enthesitis at sites where ligaments and tendons are attached to bone in structures adjacent to the hip joint (expressed as Yes or No).
Time Frame: 12 months from the baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Golimumab Injection
Number analyzed (Participants) | 18
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment (baseline) up to 2 years of follow-up during treatment.
Arm/Group | Golimumab Injection
All-Cause Mortality (participants affected / at risk) | 1/39
Serious Adverse Events (participants affected / at risk) | 3/39
Other Adverse Events (participants affected / at risk) | 12/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Golimumab Injection (N=39)
Alcohol intoxication (Injury, poisoning and procedural complications) | 1 — Fatal serious adverse event
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab Injection (N=39)
Acute respiratory viral infection (Respiratory, thoracic and mediastinal disorders) | 4 (5) — The most common AE reported
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (General disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alanine aminotransferase (ALT) level increased (Gastrointestinal disorders) | 1 (1)
Aspartate transaminase (AST) level increased (Gastrointestinal disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Pain in the breast (Reproductive system and breast disorders) | 1 (1)
Pain in metatarsophalangeal joints (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in hip joint (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain in epigastric region (Gastrointestinal disorders) | 1 (2)
Pain in gluteal region (Musculoskeletal and connective tissue disorders) | 1 (1)
Discharges from genital tract (Reproductive system and breast disorders) | 1 (1)
Itching in genital area (Skin and subcutaneous tissue disorders) | 1 (1)
Deflection of nasal septum (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colpitis (Reproductive system and breast disorders) | 1 (1)
Latent tuberculosis infection (Infections and infestations) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Mycoplasmosis (Infections and infestations) | 1 (1)
Loose stool (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Watery eyes (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Ureaplasmosis (Infections and infestations) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03557853/Prot_SAP_000.pdf